CLINICAL TRIAL: NCT06601595
Title: Spondyloarthropathy in Inflammatory Bowel Disease Patients and Evaluation of Its Response to TNF Inhibitors in Assiut University Hospital
Brief Title: Prevelance of Axial Spondylosis Arthritis in Inflammatory Bowel Disease and Its RESPONSE to Tumour Necrosis Factor (TNF) Inhibitors Treatment in Assiut University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Mohamed Nasr (Other)
Responsible Party: Sponsor-Investigator, Mohamed Nasr, Mohamednasr, Assiut University
Organization: Assiut University (Other)
Other Study IDs: SPA in IBD and response TNFI
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Disease (IBD); Spondylarthropathies; TNF-alpha Inhibitors
MeSH Terms: conditions — Inflammatory Bowel Diseases; Spondylarthropathies | interventions — Tumor Necrosis Factor Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- (TNF) inhibitors: 1- Patients taking biologic (infliximab) treatment
  Interventions: Drug: TNF inhibitors
- conventional IBD medical Treatment: patients taking conventional IBD medical Treatment
  Interventions: Drug: conventional ibd medical treatment

INTERVENTIONS:
Drug: TNF inhibitors — tumour necrosis factor inhibitors approved as treatments for ulcerative colitis and/or Crohns disease
  Groups: (TNF) inhibitors
Drug: conventional ibd medical treatment — Conventional therapies for ulcerative colitis and Crohns disease (CD) include aminosalicylates, corticosteroids, thiopurines, methotrexate other than anti-tumor necrosis factor agents.
  Groups: conventional IBD medical Treatment

SUMMARY:
Prevelance of axial spondylosis arthritis in inflammatory bowel disease and its RESPONSE to tumour necrosis factor (TNF) inhibitors TREATMENT

DETAILED DESCRIPTION:
Inflammatory bowel disease [IBD], encompassing Crohn's disease and ulcerative colitis, represents a chronic inflammatory disease entity that mainly affects the gastrointestinal tract.1 Extraintestinal manifestations, however, frequently occur and may involve different organ systems.2 Among the most common extraintestinal manifestations are spondyloarthritis [SpA], here defined as ankylosing spondylitis, psoriatic arthritis, enteropathic arthritis, reactive arthritis, and undifferentiated spondyloarthritis diagnosis.3 This group of rheumatic diseases share a similar clinical presentation with involvement of the spine, sacroiliac joints, peripheral arthritis, and frequently also enthesitis.4 Both IBD and SpA are also highly heritable diseases, and genome-wide and family-based association studies have demonstrated evidence of a shared genetic basis between IBD and SpA.5-6 Comorbidity with SpA has been associated with disability and decreased quality of life in IBD patients.7 In some IBD patients, these complications of SpA can lead to greater morbidity than the typical gastrointestinal symptoms for IBD.8 Even though lower back pain is commonly reported by IBD patients with SpA, early symptoms related to SpA may be mild and not always recognisable. However, an early diagnosis of SpA is important since a delayed diagnosis may potentially lead to a more severe disease course and poor treatment responses in patients with SpA.9 Infliximab is a genetically constructed immunoglobulin (Ig)G1 murine-human chimeric monoclonal antibody that binds the soluble subunit and the membrane-bound precursor of tumor necrosis factor-α (TNF-α). Consequently, it helps to decrease the biological activity of TNF-α (10). Neutralization of TNF-α has been suggested as a therapeutic strategy for patients with inflammatory bowel disease (IBD), rheumatoid arthritis (RA), spondyloarthropathy (SpA) and various other chronic inﬂammatory conditions (11).

ELIGIBILITY:
Inclusion Criteria:IBD patients (ulcerative colitis , Crohn's disease )on TNF inhibitors Data collected included SPA and IBD variables, demographics, concurrent medications, co-morbidities and autoimmune serology.

They fulfil criteria of axial SPA Clinical Criteria 12 Low back pain ≥ 3 months, improved by exercise and not relieved by rest Limitation of lumbar spine in sagittal and frontal planes Limitation of chest expansion (relative to normal values corrected for age and sex) Radiological Criteria Bilateral grade 2-4 sacroiliitis, or; Unilateral 3-4 sacroiliitis Assessment of disease activity of SPA 13 Patient fulfill criteria of IBD 14 Assessment of IBD activity (Esr , CRP ,Faecal calprotectin , CBC , albumin ,endoscopy, histopathology) Mayo score for U.C Crohn's disease Activity index

Exclusion Criteria: Other autoimmune disease , DM, LCF ,CRF ,Malignancy , Mechanical low back pain, Fracture , Spondylolisthesis , Spine tumores , Kidney stones .

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: IBD patients (ulcerative colitis , Crohs disease ) in gastroenterology department ,ASSUIT UNIVERSITY hospital and EL RAGHY hospital inpatient and outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
prevalence of SPA in IBD patients | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Salwa salaheldin elgendi, professor doctor, Study Director — Assiut University; hossam Mahmoud AbdulWahab, assistant professor, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Van Deventer SJ. Tumour necrosis factor and Crohn's disease. Gut. 1997 Apr;40(4):443-8. doi: 10.1136/gut.40.4.443. No abstract available. PMID 9176068
- [Result] Everhov AH, Khalili H, Askling J, Myrelid P, Ludvigsson JF, Halfvarson J, Nordenvall C, Soderling J, Olen O, Neovius M. Sick Leave and Disability Pension in Prevalent Patients With Crohn's Disease. J Crohns Colitis. 2018 Nov 28;12(12):1418-1428. doi: 10.1093/ecco-jcc/jjy123. PMID 30165593
- [Result] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Result] Hedin CRH, Vavricka SR, Stagg AJ, Schoepfer A, Raine T, Puig L, Pleyer U, Navarini A, van der Meulen-de Jong AE, Maul J, Katsanos K, Kagramanova A, Greuter T, Gonzalez-Lama Y, van Gaalen F, Ellul P, Burisch J, Bettenworth D, Becker MD, Bamias G, Rieder F. The Pathogenesis of Extraintestinal Manifestations: Implications for IBD Research, Diagnosis, and Therapy. J Crohns Colitis. 2019 Apr 26;13(5):541-554. doi: 10.1093/ecco-jcc/jjy191. PMID 30445584
- [Result] Thjodleifsson B, Geirsson AJ, Bjornsson S, Bjarnason I. A common genetic background for inflammatory bowel disease and ankylosing spondylitis: a genealogic study in Iceland. Arthritis Rheum. 2007 Aug;56(8):2633-9. doi: 10.1002/art.22812. PMID 17665420
- [Result] Lowenberg M. Anti-TNF Agents in Elderly IBD Patients: Cause for Concern? J Crohns Colitis. 2020 Jul 30;14(7):881-882. doi: 10.1093/ecco-jcc/jjaa025. No abstract available. PMID 32577750
- [Result] Beaugerie L, Rahier JF, Kirchgesner J. Predicting, Preventing, and Managing Treatment-Related Complications in Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2020 May;18(6):1324-1335.e2. doi: 10.1016/j.cgh.2020.02.009. Epub 2020 Feb 12. PMID 32059920
- [Result] Singh S, Fumery M, Sandborn WJ, Murad MH. Systematic review and network meta-analysis: first- and second-line biologic therapies for moderate-severe Crohn's disease. Aliment Pharmacol Ther. 2018 Aug;48(4):394-409. doi: 10.1111/apt.14852. Epub 2018 Jun 19. PMID 29920733
- [Result] Loftus CG, Loftus EV Jr, Harmsen WS, Zinsmeister AR, Tremaine WJ, Melton LJ 3rd, Sandborn WJ. Update on the incidence and prevalence of Crohn's disease and ulcerative colitis in Olmsted County, Minnesota, 1940-2000. Inflamm Bowel Dis. 2007 Mar;13(3):254-61. doi: 10.1002/ibd.20029. PMID 17206702
- [Result] Salvarani C, Vlachonikolis IG, van der Heijde DM, Fornaciari G, Macchioni P, Beltrami M, Olivieri I, Di Gennaro F, Politi P, Stockbrugger RW, Russel MG; European Collaborative IBD Study Group. Musculoskeletal manifestations in a population-based cohort of inflammatory bowel disease patients. Scand J Gastroenterol. 2001 Dec;36(12):1307-13. doi: 10.1080/003655201317097173. PMID 11761022